CLINICAL TRIAL: NCT02687074
Title: Effects of High Flow Nasal Canula on Moderate and Severe Respiratory Failure Patients
Brief Title: Effects of HFNC on Moderate and Severe Respiratory Failure Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Southeast University, China (Other)
Collaborators: First Affiliated Hospital of Suzhou Medical College (Other); Second Affiliated Hospital of Suzhou University (Other); Zhangjiagang First People's Hospital (Other); The Second Hospital of Nanjing Medical University (Other); Wuxi No. 4 People's Hospital (Other)
Responsible Party: Principal Investigator, Chun Pan, Principal Investigator, Southeast University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: |HFNC study
Record Dates: First submitted 2016-01-27; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Respiratory Failure
Keywords: HFNC; Respiratory Failure; Intubation; Mortality
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intubation rate on 28 days (Experimental): patients with respiratory failure treat with HFNC or NIV and intubation rate on 28 days
  Interventions: Device: HFNC; Device: NIV

INTERVENTIONS:
Device: HFNC — patients treated with high flow nasal cannula
Device: NIV — patients treated with noninvasive ventilation

SUMMARY:
Respiratory failure is the danger for the patients admitted in ICU, mechanical ventilation could save a lot of patients' life, however, it prolongs patients' ICU stay and hospital stay. High flow nasal cannula (HFNC) has advantages of PEEP effects, reducing dead space, increasing EELV and improving comfort, and it has been used to treat respiratory failure patients. In recent study, HFNC could improve mortality of respiratory failure patients with P/F<200mmHg in the subgroup. The investigators want to start a randomized controlled study to evaluate the effects of HFNC on the patients with respiratory failure.

DETAILED DESCRIPTION:
just as the brief summary

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years
2. patients met all four of the following criteria:

   * a respiratory rate of more than 25 breaths per minute,
   * a ratio of the partial pressure of arterial oxygen (Pao2) to the Fio2 of 300 mm Hg or less while the patient was breathing oxygen at a flow rate of 10 liters per minute or more for at least 15 minutes,
   * a partial pressure of arterial carbon dioxide (Paco2) not higher than 45 mmHg, and
   * an absence of clinical history of underlying chronic respiratory failure

Exclusion Criteria:

1. Paco2 of more than 45 mm Hg
2. exacerbation of asthma or chronic respiratory failure
3. cardiogenic pulmonary edema
4. severe neutropenia
5. hemodynamic instability, use of vasopressors,
6. Glasgow Coma Scale score of 12 points or less (on a scale from 3 to 15, with lower scores indicating reduced levels of consciousness)
7. contraindications to noninvasive ventilation
8. urgent need for endotracheal intubation, a do-not-intubate order, and a decision not to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
intubation rate on 28 days | up to 28 days

SECONDARY OUTCOMES:
Duration of ICU stay | date of death from any cause, whichever came first, assessed up to 90 days
Duration of hospital stay | date of death from any cause, whichever came first, assessed up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Chun Pan, Dr, Study Chair — Zhongda hospital, Southeast University, Jiangsu, China; Fuxi Sun, Dr, Principal Investigator — Nanjing Medical University affiliated Second Hospital; Wei Liu, Dr, Principal Investigator — Wuxi Hospital; Jianfeng Xie, Dr, Principal Investigator — Suzhou Shili Hospital; Songqiao Liu, Dr, Principal Investigator — Suzhou Sencond Hospital; Ling Liu, Dr, Principal Investigator — Zhangjiagang Hospital

IPD SHARING:
Plan to Share IPD: Undecided